CLINICAL TRIAL: NCT04428203
Title: A Phase I/Ib Study on the Safety of Epidiolex in Patients With Prostate Cancer With Rising PSA After Localized Therapy With Either Surgery or Radiation
Brief Title: Epidiolex (CBD) in Patients With Biochemically Recurrent Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zin W Myint (Other)
Responsible Party: Sponsor-Investigator, Zin W Myint, Assistant Professor of Medicine, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20-GU-74-PMC
Record Dates: First submitted 2020-06-06; First posted 2020-06-11 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer Recurrent; Prostate Cancer; Prostate Adenocarcinoma
Keywords: Prostate; Rising PSA; CBD Oil; Epidiolex
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation: Epidiolex 600 mg (Experimental): Cohort 1 participants with rising PSA after failure of localized therapy will receive 600 mg oral solution Epidiolex once daily for a total of 90 days in the absence of disease progression or unacceptable toxicity followed by a 10-day taper with 30 days of follow up after the discontinuation (last dose) of Epidiolex
  Interventions: Drug: Epidiolex Oral Liquid Product
- Dose Escalation: Epidiolex 800 mg (Experimental): Cohort 2 participants with rising PSA after failure of localized therapy will receive 800 mg oral solution Epidiolex once daily for a total of 90 days in the absence of disease progression or unacceptable toxicity followed by a 10-day taper with 30 days of follow up after the discontinuation (last dose) of Epidiolex
  Interventions: Drug: Epidiolex Oral Liquid Product
- Dose Expansion: Epidiolex 800 mg (Experimental): Expansion Cohort participants with rising PSA after failure of localized therapy will receive the MTD of 800 mg oral solution Epidiolex once daily for a total of 90 days in the absence of disease progression or unacceptable toxicity followed by a 10-day taper with 30 days of follow up after the discontinuation (last dose) of Epidiolexdose
  Interventions: Drug: Epidiolex Oral Liquid Product

INTERVENTIONS:
Drug: Epidiolex Oral Liquid Product — 600 mg Oral solution
  Other Names: CBD oil
  Arms: Dose Escalation: Epidiolex 600 mg
Drug: Epidiolex Oral Liquid Product — 800 mg oral solution
  Other Names: CBD oil
  Arms: Dose Escalation: Epidiolex 800 mg
Drug: Epidiolex Oral Liquid Product — 800 mg oral solution
  Other Names: CBD oil
  Arms: Dose Expansion: Epidiolex 800 mg

SUMMARY:
The purpose of this phase I/Ib study is to determine the safety profile of Epidiolex (CBD oil) in biochemically recurrent prostate cancer patients. The study consists of a dose escalation part and dose expansion part. The dose expansion part of the study will use the maximum tolerated dose (MTD) determined in the dose escalation part to assess the activity, safety and tolerability of the investigational product in patients with biochemically recurrent prostate cancer after localized therapy with either surgery or radiation.

DETAILED DESCRIPTION:
Cannabinoids (CBD) have been widely used in medicines for centuries to control pain, nausea or vomiting, and to stimulate appetite, especially in cancer patients. Both cannabinoids receptor 1(CB1) and cannabinoids receptor 2 (CB2) were highly expressed in cultured prostate cancer cells compared to normal prostate cell lines. CBD inhibits tumor growth in xenograft model.

Clinicians have been challenged to improve the treatment of biochemically recurrent (BCR) prostate cancer in which prostatic specific antigen (PSA) rises without radiological or clinical progression years after localized treatment (radical prostatectomy or radiation therapy) with or without hormonal treatment. Approximately 50-90% of men with high-risk prostate cancer will experience a BCR. Based on the abovementioned preclinical observations of CBD's effect on prostate cancer and its safety data in two non-cancer populations, a phase I study of CBD in men with biochemically recurrent prostate cancer will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Completion of localized therapy (prostatectomy or radiotherapy) for prostate adenocarcinoma (either histologically or cytologically confirmed)
* Biochemical (PSA) recurrence, defined as: * PSA of >= 0.2 ng/ml that has increased above nadir following radical prostatectomy OR * PSA increase of 2.0 ng/ml above post-therapy nadir after radiotherapy NOTE: PSA measured at two consecutive time points (separated by 4 or more weeks) is required in order to demonstrate the requisite increase in PSA
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count >= 1,500/microliters (at baseline [pre-study])
* Platelets >= 80,000/microliters (at baseline [pre-study])
* Total bilirubin =< institutional upper limit of normal (at baseline [pre-study])
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase) =< institutional upper limit of normal (at baseline [pre-study])
* Glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2 using the Cockcroft-Gault formula (at baseline [pre-study])
* Patients with a prior or concurrent malignancy (non-prostate) whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen as determined by the treating physician are eligible
* Given that worsening of an underlying state of mental depression or suicidal ideation has been reported with Epidiolex, patients should be carefully screened for depression at baseline and if there are indications or a history of depression it is strongly recommended that these patients be closely followed together with behavioral health or psychiatric medical support. Patients with an established diagnosis of depression that, in the assessment of the investigator may make the administration of Epidiolex hazardous, should not be enrolled on this protocol
* Concurrent use of over-the-counter CBD oil, Marinol or marijuana is not permitted. Patients with a history of current over-the-counter CBD oil, Marinol or marijuana use for any reason are eligible only if they do the following: * Complete a one-week washout period prior to study initiation * Refrain from non-study related CBD oil, Marinol or marijuana use while on-study
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of hypersensitivity to Epidiolex (cannabidiol) or sesame seeds (one of the inactive ingredients in Epidiolex)
* Any radiological evidence of metastatic disease (determined by standard of care computed tomography [CT] scans of abdomen. pelvis, chest, whole body bone scan or Axium positron emission tomography scan). Questionable lesions on bone scan will be confirmed by standard of care methods such as plain X-rays or Axium positron emission tomography scan, if not previously performed
* Receipt of prior cytotoxic chemotherapy for recurrent prostate cancer
* Use of androgen deprivation therapy (for example, bicalutamide, flutamide, nilutamide, or leuprolide acetate) concurrently or within the previous 3 months.
* Uncontrolled intercurrent illness such as active infections. Other illnesses will be evaluated and eligibility status determined at the discretion of the treating physician and the investigator
* Psychiatric illness/social situations that would limit compliance with study requirements
* Concomitant use of valproate or clobazam
* Concurrent use of over-the-counter CBD oil, Marinol or marijuana
* Epidiolex is a moderate inhibitor of CYP2C19 and a moderate/strong inhibitor of CYP3A4, therefore concurrent use of CYP2C19 substrates is not allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate cancer only occurs in male
Enrollment: 21 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zin W. Myint, MD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Dose Escalation: Epidiolex 600 mg: Cohort 1 participants with rising PSA after failure of localized therapy will receive 600 mg oral solution Epidiolex once daily for a total of 90 days in the absence of disease progression or unacceptable toxicity followed by a 10-day taper with 30 days of follow up after the discontinuation (last dose) of Epidiolex
- Experimental: Dose Escalation: Epidiolex 800 mg: Cohort 2 participants with rising PSA after failure of localized therapy will receive 800 mg oral solution Epidiolex once daily for a total of 90 days in the absence of disease progression or unacceptable toxicity followed by a 10-day taper with 30 days of follow up after the discontinuation (last dose) of Epidiolex
- Experimental: Dose Expansion: Epidiolex 800 mg: Expansion Cohort participants with rising PSA after failure of localized therapy will receive the MTD of 800 mg oral solution Epidiolex once daily for a total of 90 days in the absence of disease progression or unacceptable toxicity followed by a 10-day taper with 30 days of follow up after the discontinuation (last dose) of Epidiolexdose
Period: Overall Study
Arm/Group | Experimental: Dose Escalation: Epidiolex 600 mg | Experimental: Dose Escalation: Epidiolex 800 mg | Experimental: Dose Expansion: Epidiolex 800 mg
Started | 4 | 3 | 14
Completed | 2 | 3 | 13
Not Completed | 2 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dose Escalation and Dose Expansion: Epidiolex 800 mg: Cohort 2 participants with rising PSA after failure of localized therapy will receive 800 mg oral solution Epidiolex once daily for a total of 90 days in the absence of disease progression or unacceptable toxicity followed by a 10-day taper with 30 days of follow up after the discontinuation (last dose) of Epidiolex Expansion Cohort participants with rising PSA after failure of localized therapy will receive the MTD of 800 mg oral solution Epidiolex once daily for a total of 90 days in the absence of disease progression or unacceptable toxicity followed by a 10-day taper with 30 days of follow up after the discontinuation (last dose) of Epidiolexdose
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: Epidiolex 600 mg | Dose Escalation and Dose Expansion: Epidiolex 800 mg | Total
Number analyzed (Participants) | 4 | 17 | 21
Age, Continuous [Median (Full Range); unit: years] | 68 [66 to 72] | 71 [47 to 85] | 69 [47 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 17 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 3 | 14 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 17 | 21
PSA (ng/ml) [Median (Full Range); unit: ng/ml] | 1.84 [0.41 to 6.12] | 1.25 [0.24 to 16.3] | 1.25 [0.24 to 16.3]
Testosterone, total (ng/dL) [Median (Full Range); unit: mg/dL] | 214.5 [7 to 505] | 360 [142 to 1166] | 325 [7 to 1166]
Prior treatment [Count of Participants; unit: Participants]
  Prostatectomy Alone | 1 | 3 | 4
  Radiation Alone | 1 | 4 | 5
  Prostatectomy and salvage radiation | 2 | 10 | 12
  Untreated | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (Treatment-related Adverse Events) as Assessed by the CTCAE v5.0
Description: DLT was defined as grade ≥3 nausea, vomiting, diarrhea that persists >72 h despite optimal anti-emetics and anti-diarrhea treatment, grade ≥3 hematological adverse events (AEs), or grade ≥2 suicidal ideation.Treatment-related adverse events are those that comprise a dose-limiting toxicity within 30 days after initiation of Epidiolex (i.e., acute DLT). Additionally, Treatment-related adverse events will continue to be monitored for a total of 90 days.
Time Frame: up to 90 days
Population: Among 21 patients, a total of 18 patients were included in the efficacy analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Epidiolex 600 mg | Dose Escalation: Epidiolex 800 mg | Dose Expansion: Epidiolex 800 mg
Number analyzed (Participants) | 2 | 3 | 13
Participants | 0 | 0 | 0

2. Secondary Outcome: Participants With Biochemical Response.
Description: Biochemical response (25% change from baseline) will be determined by the measurement of PSA at baseline and approximately every 4 weeks during treatment.
Time Frame: within 90 days
Population: Patients who were DLT evaluable, had baseline measurements, and had at least one post-baseline measurement were included in the analysis of secondary endpoints. The assessments were combined for patients who received the recommended dose of 800 mg daily.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation and Expansion: Epidiolex 800 mg: Both Escalation and Expansion Cohorts participants with rising PSA after failure of localized therapy will receive the MTD of 800 mg oral solution Epidiolex once daily for a total of 90 days in the absence of disease progression or unacceptable toxicity followed by a 10-day taper with 30 days of follow up after the discontinuation (last dose) of Epidiolexdose
Arm/Group | Dose Escalation: Epidiolex 600 mg | Dose Escalation and Expansion: Epidiolex 800 mg
Number analyzed (Participants) | 2 | 16
Participants
  stable biochemical disease | 2 | 14
  partial biochemical response | 0 | 1
  PSA progression | 0 | 1

3. Secondary Outcome: Change in PSA Velocity From Baseline Throughout the Treatment Period as an Indication of Biochemical Response.
Description: Biochemical response will be determined by measurement of PSA approximately every 4 weeks during treatment. PSA velocity is the calculation (PSA final measurement - PSA initial measurement) / number of years between measurements.
Time Frame: within 90 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanograms per milliliter per year
Arm/Group | Dose Escalation and Expansion: Epidiolex 800 mg | Dose Escalation: Epidiolex 600 mg
Number analyzed (Participants) | 16 | 2
nanograms per milliliter per year | 0 (0) | 0 (0)

4. Secondary Outcome: Change in Testosterone Levels From Baseline Throughout the Treatment Period as an Indication of Biochemical Response
Description: Biochemical response will be determined by measurement of total testosterone level approximately every 4 weeks during treatment.
Time Frame: Baseline, Day 1 of Cycle 1 (each cycle is 4 weeks), Day 1 of Cycle 2, Day 1 of Cycle 3, and 1 month post treatment (up to 16 weeks)
Population: Patients who were DLT evaluable, had baseline measurements, and had at least one post-baseline measurement were included in the analysis of secondary endpoints. Data analysis for this outcome was combined in the 800 mg group
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Dose Escalation and Expansion: Epidiolex 800 mg | Dose Escalation: Epidiolex 600 mg
Number analyzed (Participants) | 16 | 2
ng/dL
  Baseline: number analyzed (Participants) | 15 | 2
  Baseline | 388.3 (270.7) | 214.5 (30.4)
  Cycle 1 | 421.94 (238.67) | 190 (76.37)
  Cycle 2: number analyzed (Participants) | 14 | 2
  Cycle 2 | 345.21 (157.02) | 242 (14.14)
  Cycle 3: number analyzed (Participants) | 12 | 2
  Cycle 3 | 253.92 (249.61) | 208 (36.77)
  1 month post treatment | 434.0 (252.8) | 190.0 (76.4)

5. Secondary Outcome: Health-related Quality of Life (EORTC Quality of Life Questionnaire-C30)
Description: The EORTC quality of life questionnaire (QLQ) 30 is a validated 30-item patient-reported questionnaire assessing quality of life among cancer populations. The quality of life questionnaire-C30 is the core QOL instrument, with 30 items that comprise five functioning scales (physical, social, role, cognitive, and emotional functioning), eight symptom scales (fatigue, nausea/vomiting, pain, dyspnea, sleep disturbances, appetite loss, constipation, and diarrhea), financial impact, and overall quality of life. All raw item scores are transformed to scale scores, linearly converted to range from 0 to 100. For the functioning scales and global QOL, higher scores indicate better functioning. For the symptom scales, higher scores indicate higher symptom burden.
Time Frame: Baseline
Population: No data released for 600mg as only 1 participant answered QOL measures and confidentiality of health information could be impacted if the outcome measures were displayed. Only patients who received one or more doses of the recommended phase 2 dose (800 mg) and who completed one or more sections of the quality-of-life assessment were analyzed. Of the 17 patients who received the recommended dose of 800 mg daily, 17 completed patient-reported outcomes at baseline and 12 completed PROs at 12 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dose Escalation and Expansion: Epidiolex 800 mg | Dose Escalation: Epidiolex 600 mg
Number analyzed (Participants) | 17 | 0
units on a scale
  Global Health Status/QOL | 78.4 (15.0) |
  Physical Functioning | 92.9 (11.9) |
  Role Functioning | 97.1 (8.8) |
  Emotional Functioning | 94.1 (9.2) |
  Cognitive Functioning | 93.1 (10.3) |
  Social Funcitoning | 97.1 (8.8) |
  Fatigue | 12.4 (13.0) |
  Nausea/Vomiting | 1.0 (4.0) |
  Pain | 15.7 (21.6) |
  Dyspnea | 7.8 (14.6) |
  Insomnia | 13.7 (16.9) |
  Appetite Loss | 0.0 (0.0) |
  Constipation | 3.9 (11.1) |
  Diarrhea | 7.8 (14.6) |
  Financial Problems | 7.8 (14.6) |

6. Secondary Outcome: Health-related Quality of Life (EORTC Quality of Life Questionnaire-C30)
Description: as for outcome 5
Time Frame: 12 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dose Escalation and Expansion: Epidiolex 800 mg | Dose Escalation: Epidiolex 600 mg
Number analyzed (Participants) | 12 | 0
units on a scale
  Global Health Status/QOL | 81.3 (13.4) |
  Physical Functioning | 90.0 (14.4) |
  Role Functioning | 93.1 (13.2) |
  Emotional Functioning | 96.5 (5.6) |
  Cognitive Functioning | 91.7 (11.2) |
  Social Funcitoning | 95.8 (10.4) |
  Fatigue | 16.7 (18.7) |
  Nausea/Vomiting | 1.4 (4.8) |
  Pain | 13.9 (17.2) |
  Dyspnea | 13.9 (22.3) |
  Insomnia | 8.3 (20.7) |
  Appetite Loss | 0.0 (0.0) |
  Constipation | 13.9 (17.2) |
  Diarrhea | 8.3 (15.1) |
  Financial Problems | 11.1 (16.4) |

7. Secondary Outcome: Prostate Cancer-Specific Quality of Life (EORTC Quality of Life Questionnaire-PR25)
Description: The EORTC quality of life questionnaire (QLQ)-PR25 is a validated 25-item patient-reported questionnaire which complements the EORTC QLQ-C30,core QOL questionnaire. The QLQ-PR25 comprises 25 items assessing sequelae specific to prostate cancer and its treatment, and thus, is intended to supplement the EORTC QLQ-C30. The 25 items comprise six prostate-specific scales: Urinary, Bowel, Use of Incontinence Aids, Prostate Cancer Treatment-Related Symptoms, Sexual Active and Sexual Function. Raw item scores are linearly transformed to a 0 to 100 scale (i.e., same unit of measurement used by the core QLQ-C30 questionnaire). For the QLQ-PR25, higher scores on symptom domains (e.g., urinary, bowel, etc.) indicate greater symptom burden. Higher scores on function domains (e.g., Sexual Function) indicate better functioning.
Time Frame: Baseline
Population: Assessments were combined and analyzed for patients who received one or more doses of the recommended phase 2 dose and who completed one or more sections of the quality-of-life assessment. For 800mg dose17 completed baseline and 12 completed at 12 weeks. Some participants left some questions blank (incontinence, sexual activity). No data released for 600mg as only 1 participant answered QOL measures, confidentiality of health information could be impacted if the outcome measures were displayed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dose Escalation and Expansion: Epidiolex 800 mg | Dose Escalation: Epidiolex 600 mg
Number analyzed (Participants) | 17 | 0
units on a scale
  Urinary Symptoms | 17.9 (12.7) |
  Incontinence aid: number analyzed (Participants) | 7 | 0
  Incontinence aid | 9.5 (16.3) |
  Bowel Symptoms | 6.4 (8.1) |
  Hormonal Treatment Related Symptoms | 5.9 (6.0) |
  Sexual activity | 67.6 (22.3) |
  Sexual Functioning: number analyzed (Participants) | 8 | 0
  Sexual Functioning | 56.9 (26.8) |

8. Secondary Outcome: Prostate Cancer-Specific Quality of Life (EORTC Quality of Life Questionnaire-PR25)
Description: as for outcome 7
Time Frame: 12 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dose Escalation and Expansion: Epidiolex 800 mg | Dose Escalation: Epidiolex 600 mg
Number analyzed (Participants) | 12 | 0
units on a scale
  Urinary Symptoms | 17.5 (11.2) |
  Incontinence aid: number analyzed (Participants) | 3 | 0
  Incontinence aid | 22.2 (19.2) |
  Bowel Symptoms | 7.6 (8.3) |
  Hormonal Treatment Related Symptoms | 9.0 (10.2) |
  Sexual activity | 63.9 (21.1) |
  Sexual Functioning: number analyzed (Participants) | 2 | 0
  Sexual Functioning | 77.8 (0.0) |

ADVERSE EVENTS:
Time Frame: 120 days
Description: Toxicities were graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Groups:
- Experimental: Dose Escalation and Expansion: Epidiolex 800 mg: Both Escalation and Expansion Cohorts participants with rising PSA after failure of localized therapy will receive the MTD of 800 mg oral solution Epidiolex once daily for a total of 90 days in the absence of disease progression or unacceptable toxicity followed by a 10-day taper with 30 days of follow up after the discontinuation (last dose) of Epidiolexdose
Arm/Group | Experimental: Dose Escalation: Epidiolex 600 mg | Experimental: Dose Escalation and Expansion: Epidiolex 800 mg
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/17
Other Adverse Events (participants affected / at risk) | 2/2 | 9/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Dose Escalation: Epidiolex 600 mg (N=2) | Experimental: Dose Escalation and Expansion: Epidiolex 800 mg (N=17)
Diarrhea (Gastrointestinal disorders) | 2 | 9
Nausea (Gastrointestinal disorders) | 2 | 3
Bloating (Gastrointestinal disorders) | 0 | 1
Stomach Pain (Gastrointestinal disorders) | 0 | 1
Abnormal Liver Function Test (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 2 | 2
Malaise (General disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Insomnia (Nervous system disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT04428203/Prot_SAP_ICF_001.pdf